CLINICAL TRIAL: NCT07394439
Title: Association of Respiratory Function and Respiratory Muscle Strength With Hand Function in Children With Hemiparetic Cerebral Palsy
Brief Title: Respiratory Function, Respiratory Muscle Strength, and Hand Function in Hemiparetic Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, İrem Çetinkaya, Assistant Professor, Halic University
Other Study IDs: Acetinkaya009
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Palsy; Respiratory Function Tests; Fine Motor Skills
Keywords: Hemiparetic Cerebral Palsy; Respiratory Function; Respiratory Muscle Strength; Hand Function
MeSH Terms: conditions — Cerebral Palsy; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn how respiratory function and respiratory muscle strength are related to hand use in children and teenagers with hemiparetic cerebral palsy (CP) aged 6 to 18 years.

The main questions it aims to answer are:

Is respiratory function related to hand function in children with hemiparetic CP? Is respiratory muscle strength related to hand function in children with hemiparetic CP? Is respiratory function related to how strong children can squeeze with their affected hand? Is respiratory muscle strength related to how strong children can squeeze with their affected hand? Is respiratory function related to how well children use their hands in daily activities? Is respiratory muscle strength related to how well children use their hands in daily activities? Is respiratory function related to children's hand skill level? Is respiratory muscle strength related to children's hand skill level?

Participants will:

Visit the clinic one time for a single assessment session. Do simple lung tests using a small portable device to measure respiratory function.

Do tests that measure how strong their breathing muscles are.

Complete hand and arm tests, including:

A hand grip strength test, A simple block-moving test, A short questionnaire about using the hand in daily life, A standard hand skill rating. Researchers will look at how respiratory measures are related to hand strength, hand skills, and daily hand use. This study may help improve rehabilitation programs by showing whether respiratory muscle strength and hand skills should be trained together in children with hemiparetic CP.

DETAILED DESCRIPTION:
Hemiparetic cerebral palsy (CP) is associated with asymmetric motor impairments that may affect trunk stability, respiratory mechanics, and hand function. This observational, cross-sectional study aims to examine the relationship between respiratory function, respiratory muscle strength, and hand function in children with hemiparetic CP.

The study will include at least 37 participants aged 6 to 18 years with a diagnosis of hemiparetic CP. Demographic and clinical characteristics will be recorded. Respiratory function will be assessed using a portable spirometer, and respiratory muscle strength will be measured by maximum inspiratory and expiratory pressures. Hand function will be evaluated using grip strength (Jamar dynamometer), gross manual dexterity (Box and Block Test), functional hand use in daily activities (ABILHAND-Kids), and manual ability level (MACS).

All assessments will be conducted in a single session under standardized conditions by the same physiotherapist. Data will be analyzed using descriptive statistics and Pearson or Spearman correlation tests. Comparisons between different functional levels will also be performed.

The findings are expected to clarify the interaction between respiratory capacity and upper extremity function and to support comprehensive rehabilitation approaches targeting both hand skills and respiratory muscle strength in children with hemiparetic CP.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hemiparetic cerebral palsy by a physician.
* Sufficient cognitive ability to understand and follow test instructions, as judged by a parent or clinician.
* Clinically stable condition for at least 3 months, with no changes in medication, acute exacerbations, or modifications in rehabilitation programs.
* Physical capacity sufficient to tolerate pulmonary function testing (spirometry), maximum inspiratory/expiratory pressure (MIP/MEP) measurements, and other study assessments.

Exclusion Criteria:

* Current or recent acute respiratory infection, asthma exacerbation, pneumonia, or known cardiopulmonary disease that may affect testing.
* Receipt of intensive upper extremity interventions other than routine physiotherapy (e.g., botulinum toxin injections, surgical procedures) within the past 6 months.
* History of major orthopedic surgery (e.g., hip reconstruction, scoliosis surgery) within the past 3 months.
* Severe musculoskeletal contracture or deformity that prevents the safe performance of pulmonary function testing.
* Severe epilepsy, uncontrolled seizures, or other neurological conditions that may compromise safety during testing.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 6-18 years with a physician-confirmed diagnosis of hemiparetic cerebral palsy, recruited from outpatient pediatric rehabilitation clinics and physiotherapy centers. Participants will be individuals receiving routine follow-up or rehabilitation services who meet the study eligibility criteria and are able to complete respiratory and hand function assessments.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure | Baseline (single assessment session)
  Respiratory muscle strength related to inspiration will be assessed in accordance with the joint recommendations of the American Thoracic Society and the European Respiratory Society. Measurements will be performed using a portable electronic respiratory pressure device (Cosmed Pony Fx, Rome, Italy). Participants will wear a mouthpiece and a nose clip to prevent air leakage. After full expiration, participants will perform a maximal inspiratory effort. The measurement will be repeated three times, and the highest value will be recorded for analysis.
  Outcome Measure Units cmH2O
Maximum Expiratory Pressure | Baseline (single assessment session)
  Respiratory muscle strength related to expiration will be assessed in accordance with the joint recommendations of the American Thoracic Society and the European Respiratory Society. Measurements will be performed using the same portable electronic respiratory pressure device. Participants will wear a mouthpiece and a nose clip to prevent air leakage. After full inspiration, participants will perform a maximal expiratory effort. The measurement will be repeated three times, and the highest value will be recorded for analysis.
  Outcome Measure Units cmH2O
Forced Vital Capacity | Baseline (single assessment session)
  Pulmonary function will be assessed by spirometry in accordance with the standards of the American Thoracic Society and the European Respiratory Society using a portable spirometer (COSMED Pony Fx, Rome, Italy). Measurements will be performed in a seated position with back support while participants wear a nose clip. Participants will take a maximal inspiration followed by a forceful, maximal expiration. Three trials will be performed, and the highest acceptable value will be recorded for analysis.
  Unit of Measure liters
Forced Expiratory Volume in One Second | Baseline (single assessment session)
  Pulmonary function will be assessed using the same spirometry procedure and equipment. The volume of air exhaled during the first second of a forced expiration will be recorded. Three trials will be performed, and the highest acceptable value will be used for analysis.
  Unit of Measure liters
Ratio of Forced Expiratory Volume in One Second to Forced Vital Capacity Ratio | Baseline (single assessment session)
  Pulmonary function will be assessed using the same spirometry procedure and equipment. The ratio between the forced expiratory volume in one second and the forced vital capacity will be calculated from the best acceptable maneuver and recorded for analysis.
  Unit of Measure percent
Peak Expiratory Flow Rate | Baseline (single assessment session)
  Pulmonary function will be assessed using the same spirometry procedure and equipment. The highest expiratory flow achieved during the forced expiration maneuver will be recorded. Three trials will be performed, and the highest acceptable value will be used for analysis.
  Unit of Measure liters per second
Classification Level on the Manual Ability Classification System | Baseline (single assessment session)
  Manual ability will be classified using the Manual Ability Classification System (MACS), a five-level classification system that describes how children with cerebral palsy use their hands during daily activities.
  Level I represents the most independent hand use. Level V represents the most severe limitation in manual ability. The MACS is applicable to children aged 4 to 18 years and has been validated in Turkish (Cansoy et al., 2014). In this study, MACS will be used to determine the participant's baseline level of manual ability.

SECONDARY OUTCOMES:
Score on the ABILHAND-Kids Questionnaire | Baseline (single assessment session)
  Functional use of the hand in daily activities will be assessed using the ABILHAND-Kids questionnaire, a parent-reported scale developed for children aged 6 to 15 years. The scale consists of 21 items, each rated as "easy," "difficult," or "impossible" based on the child's ability to perform bimanual daily activities.
  The scale is based on Rasch analysis and specifically designed for use in children with cerebral palsy. A validated Turkish version is available, and permission for its use has been requested.
Number of Blocks Transferred in Sixty Seconds During the Box and Block Test | Baseline (single assessment session)
  Gross manual dexterity will be assessed using the Box and Block Test (BBT), a widely used measure of upper extremity gross manual function in both pediatric and adult populations. The test evaluates basic components of manual dexterity, including grasping, holding, transferring, and releasing objects.
  The BBT consists of a wooden box (53.7 × 25.4 × 8.5 cm) divided into two equal compartments by a partition, with 150 wooden cubes (2.5 cm per side) placed in one compartment. Participants will be instructed to transfer as many blocks as possible from one compartment to the other within 60 seconds. The number of blocks transferred will be counted by the examiner using a stopwatch.
  The test will be administered separately for each hand, and the total number of blocks transferred in 60 seconds will be recorded for analysis.
Classification Level on the Gross Motor Function Classification System | Baseline (single assessment session)
  Gross motor function level will be classified using the Gross Motor Function Classification System (GMFCS), an internationally accepted five-level system that describes the gross motor abilities and level of independence of children with cerebral palsy.
  Level I: Walks without limitations. Level II: Walks with limitations. Level III: Walks using a hand-held mobility device. Level IV: Self-mobility with limitations; may use powered mobility. Level V: Transported in a manual wheelchair.
Mean Hand Grip Strength of the Affected Hand Measured With a Hand Dynamometer | Baseline (single assessment session)
  Grip strength of the affected hand will be measured using a Jamar hand dynamometer, which is considered the gold standard for grip strength assessment and is recommended by the American Society of Hand Therapists.
  Participants will be seated with:
  Shoulder in adduction, Elbow flexed at 90°, Forearm in neutral position, Wrist in neutral alignment. The affected hand will be tested three times, and the mean of the three trials will be used for analysis.
  Outcome Measure Units: Kilograms

CONTACTS AND LOCATIONS:
Overall Officials: İrem Çetinkaya, PhD, Principal Investigator — Haliç University

IPD SHARING:
Plan to Share IPD: No